CLINICAL TRIAL: NCT03334201
Title: Age-associated Arterial Dysfunction, Western Diet, and Aerobic Exercise: Role of the Gut Microbiome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Douglas Seals, Distinguished Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-0633
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Aging
MeSH Terms: interventions — Diet, Western

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind crossover
Who Masked: Investigator
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western diet first (Other): To receive Western diet controlled feeding first, followed by non-Western diet controlled feeding
  Interventions: Other: Western Diet; Other: Non-Western Diet
- Non-Western diet first (Other): To receive non-Western diet controlled feeding first, followed by Western diet controlled feeding
  Interventions: Other: Western Diet; Other: Non-Western Diet

INTERVENTIONS:
Other: Western Diet — high fat (40%), high sugar (25%) and low fiber (15g/day)
Other: Non-Western Diet — low fat (25%), low sugar (15%), high fiber (30g/day)

SUMMARY:
The risk of developing cardiovascular diseases increases with aging largely due to age-related declines in the function of arteries (arterial dysfunction), which are influenced by common lifestyle factors such as consumption of a "Western" diet and lack of sufficient physical activity; thus, it is important to study how these factors interact to affect artery function. This study will determine whether changes to the gut microbiome (the collection of bacteria and other "microbes" living in the intestinal tract) with aging, Western diet consumption and aerobic exercise influence arterial function, and the biological pathways (mechanisms) involved. Specifically, the investigators will perform a randomized, single-blind, controlled feeding crossover study design (comparing Western diet to non-Western diet consumption) in young and older, exercising and non-exercising healthy adults to determine the time course effects (temporal association) of diet on the gut microbiome and arterial function. Overall, this research has potential to establish the gut microbiome as a possible target for treating/preventing age-related arterial dysfunction and reducing the risk of age-associated cardiovascular diseases.

DETAILED DESCRIPTION:
In order to investigate how age-related changes to the gut microbiome, as modulated by Western diet and exercise, influences arterial function in humans, the investigators will capitalize on the plasticity of the gut microbiome to dietary perturbations. A randomized, single-blind, 2x1-week dietary intervention crossover study (with 3 week washout) will be conducted in young (18-29 years) and old (60-79 years), exercising and non-exercising, male and female adults from all races and ethnic backgrounds. Testing will take place on the University of Colorado Boulder main campus at the Clinical and Translational Research Center (CTRC - located in the Wardenburg Health Center). Subjects will undergo telephone and in-person CTRC screening, with those eligible assigned to either Group A or Group B using block randomization stratified by age and exercise status. Group A will undergo isocaloric WD feeding (high fat [40%], high sugar [25%], low fiber [15g], low nutrient) during Phase 1 (first 1-week treatment period) and non-WD feeding (low-fat [25%], low sugar [15%], high fiber [22g], high nutrient) during Phase 2 (second 1-week treatment period). Group B will undergo the dietary interventions in the opposite order. Phases 1 and 2 will be separated by a 3-week washout period to prevent carry over effects. During each 1-week intervention period, fecal swabs will be collected daily to characterize the gut microbiome and vascular function, will be measured at baseline and after 2 and 7 days of controlled feeding to gain insight into the temporal relation between these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-29 or 60-79 years
* Participating in < 30 min aerobic exercise < 2x/wk for >3 years OR > 45 min vigorous aerobic exercise > 4x/wk for > 3 yrs
* Currently consuming levels of dietary fat intake with the 40th-60th percentile of Americans based on the NHANES survey (29-37% calories from fat)
* Healthy (no clinical disease)
* Body mass index < 30 kg/m2
* Ankle-brachial blood pressure index > 0.9
* Total cholesterol < 240 mg/dl
* Fasting plasma glucose < 110 mg/dl
* Weight stable in the past 6 months

Exclusion Criteria:

* Current or past (within 3 months of screening) use of dietary supplements, anti-inflammatory medications, drugs known to affect the gut microbiome (antibiotics, pre/probiotics, antifungals, antivirals, antiparasitics), or gastrointestinal-targeted drugs (proton pump inhibitors, H2 receptor antagonists, laxatives, antidiarrheal medications)
* Current of past (within 5 years) smoking
* Major change in health status in the last 6 months
* Chronic clinical diseases (e.g., inflammatory bowl diseases, cardiovascular disease, diabetes, neurological disorders, dementia or other brain diseases of aging)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the gut microbiome | 7 days
  Sterile fecal swabs will be collected and analyzed using 16S rRNA sequencing
Change in endothelial function | 7 days
  Brachial artery flow-mediated dilation
Change in arterial stiffness | 7 days
  Carotid-femoral pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Seals, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided